CLINICAL TRIAL: NCT02597400
Title: A Phase 1, Open-Label, Sequential, Multiple-Dose, Drug-Drug Interaction Study of Glucokinase (GK) Activator HMS5552 and Metformin in Patients With Type 2 Diabetes Mellitus (T2DM)
Brief Title: Drug-Drug Interaction Study of Glucokinase Activator HMS5552 and Metformin in T2DM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hua Medicine Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMM0104
Record Dates: First submitted 2015-10-18; First posted 2015-11-05 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Dorzagliatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HMS5552 and Metformin (Experimental): All subjects will receive the following:
  * Metformin500 mg BID on Days 1-2, only the morning dose on Day 3. Metformin will be taken 30 minutes prior to meals;
  * Metformin 500 mg BID and HMS5552 50 mg BID on Days 4-7, only the morning dose on Day 8. Metformin and HMS5552 will be taken 30 minutes prior to meals;
  * HMS5552 50 mg BID on Days 9 -12, only the morning dose on Day 13. HMS5552 will be taken 30 minutes prior to meals.
  Interventions: Drug: Metformin; Drug: HMS5552

INTERVENTIONS:
Drug: Metformin — * Metformin500 mg BID on Days 1-2, only the morning dose on Day 3. Metformin will be taken 30 minutes prior to meals;
  * Metformin 500 mg BID and HMS5552 50 mg BID on Days 4-7, only the morning dose on Day 8. Metformin and HMS5552 will be taken 30 minutes prior to meals
  Other Names: Glucophage®
Drug: HMS5552 — * Metformin 500 mg BID and HMS5552 50 mg BID on Days 4-7, only the morning dose on Day 8. Metformin and HMS5552 will be taken 30 minutes prior to meals;
  * HMS5552 50 mg BID on Days 9 -12, only the morning dose on Day 13. HMS5552 will be taken 30 minutes prior to meals.
  Other Names: GKA

SUMMARY:
This is a Phase 1, open-label, sequential, multiple-dose, drug-drug interaction study of GK activator HMS5552 and metformin in patients with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
This is a Phase 1, open-label, sequential, multiple-dose, drug-drug interaction study of GK activator HMS5552 and metformin in patients with type 2 diabetes mellitus (T2DM). The study is to assess the potential pharmacokinetic interaction between HMS5552 and metformin in subjects with T2DM. The study is also to evaluate the safety and tolerability of HMS5552 with simultaneous administration of metformin in subjects with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects between the ages of 18 and 70 years
* Body Mass Index (BMI) of approximately 22 to 38kg/m2
* HbA1c ≥7% and ≤12%
* Are capable of giving informed consent and complying with study procedures

Exclusion Criteria:

* fasting blood glucose ≤110 or ≥270mg/dL
* Type 1 diabetes mellitus, or latent autoimmune diabetes in adults
* History or symptoms of clinically significant cardiovascular disease, particularly coronary artery disease, arrhythmias, atrial tachycardia, or congestive heart disease within one year of screening
* History of liver disease and clinically significant renal disease
* Known hypersensitivity to metformin hydrochloride;
* Positive pregnancy test result;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The primary pharmacokinetics parameters of Cmax To assess the potential pharmacokinetic interaction between HMS5552 and metformin in subjects with T2DM | 13 days
  HMS5552 and metformin PK parameters: PK parameters (Cmax) will be computed for each subject per day with non-compartmental methods using the actual sampling times. Descriptive statistics will be calculated for the PK parameters per day (Days 3, 8 and 13).
  The effect of metformin on the exposure of HMS5552 will be determined by a PK comparison between the exposure of HMS5552 on Day 13 vs. on Day 8. The effect of HMS5552 on the exposure of metformin will be determined by a PK comparison between the exposure of metformin on Day 8 vs. on Day 3.

SECONDARY OUTCOMES:
The pharmacokinetics parameters of Tmax To assess the potential pharmacokinetic interaction between HMS5552 and metformin in subjects with T2DM | 13 days
  HMS5552 and metformin PK parameters: PK parameters ( Tmax) will be computed for each subject per day with non-compartmental methods using the actual sampling times. Descriptive statistics will be calculated for the PK parameters per day (Days 3, 8 and 13).
  The effect of metformin on the exposure of HMS5552 will be determined by a PK comparison between the exposure of HMS5552 on Day 13 vs. on Day 8. The effect of HMS5552 on the exposure of metformin will be determined by a PK comparison between the exposure of metformin on Day 8 vs. on Day 3.
The pharmacokinetics parameters of AUC0-24hr To assess the potential pharmacokinetic interaction between HMS5552 and metformin in subjects with T2DM | 13 days
  HMS5552 and metformin PK parameters: PK parameters (AUC0-24hr) will be computed for each subject per day with non-compartmental methods using the actual sampling times. Descriptive statistics will be calculated for the PK parameters per day (Days 3, 8 and 13).
  The effect of metformin on the exposure of HMS5552 will be determined by a PK comparison between the exposure of HMS5552 on Day 13 vs. on Day 8. The effect of HMS5552 on the exposure of metformin will be determined by a PK comparison between the exposure of metformin on Day 8 vs. on Day 3.
Safety assessments includes monitoring of adverse events (AEs), vital signs (blood pressure, pulse rate, respiratory rate and oral temperature), clinical laboratory findings, resting 12-lead electrocardiograms (ECGs), and physical examination findings. | 13 days
  Safety assessments will include monitoring of adverse events (AEs), blood glucose via glucometer readings, vital signs (blood pressure, pulse rate, respiratory rate and oral temperature), clinical laboratory findings, resting 12-lead electrocardiograms (ECGs), and physical examination findings on Day 13 , Day 8 and Day-1
Pharmacodynamic responses (serum levels) of glucose, insulin and C-peptide will be evaluated. | 13 days

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Tracey, MD, Principal Investigator — Frontage Clinical Services, Inc.
Locations (1):
- Frontage Clinical Services Inc., Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No